CLINICAL TRIAL: NCT00165620
Title: A Randomized, Open, Parallel, Optimal Injection Rate-Finding Study for E7337 in Dynamic CT of the Liver in Patients With Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E7337-J081-141
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Lesion

INTERVENTIONS:
Drug: Iomeprole

SUMMARY:
To establish the optimum injection rate for E7337 (Iomeron 350) in dynamic CT in patients who have hepatic lesions.The primary endpoint for efficacy is the contrast enhancement effect in the early arterial phase, and the primary safety endpoints are warming sensation and vascular pain.

ELIGIBILITY:
Inclusion Criteira:

* Patients scheduled for a dynamic CT scan of the liver who have at least one hepatic lesion that has been confirmed by diagnostic imaging (ultrasonography, etc.) between 1 and 35 days before the start of the study treatment.
* Patients who are 20 years or older at the time of obtaining informed consent.

Exclusion Criteria

* Items that may affect the safety evaluation of E7337

  1. Patients who have undergone or are scheduled to undergo an examination using another contrast agent between 7 days before administration of E7337 and the time of follow-up examinations on Day 8 after administration.
  2. Patients for whom follow-ups seem to be difficult to conduct until the time of examination on Day 8 (i.e. when it may fail to evaluate delayed adverse drug reactions).
  3. Patients who have undergone or are scheduled to undergo surgical treatment or a therapy such as percutaneous ethanol injection therapy, percutaneous microwave coagulation therapy, radiofrequency ablation, or transcatheter arterial embolization, etc., from the time diagnostic imaging such as abdominal ultrasonography is performed up until follow-up examinations are conducted on Day 8 after administration.
  4. Patients who continuously need to take analgesics between the morning of administration of E7337 and the completion of CT examinations.
  5. Patients who are currently participating in another clinical study.
  6. Patients who participated in another clinical study within 3 months prior to providing informed consent for this study.
  7. Patients weighing less than 55 kg (body weight at the time of obtaining informed consent).
* General concerns relating to the safety of the subject.

  1. Patients in the acute stage with clinically unstable symptoms, or in a life-threatening condition (when it is expected that emergency treatment is required between the time of registration and the end of the follow-up period, or when the patient is not expected to survive for 3 months following administration of E7337, etc.)
  2. Patients with a history of hypersensitivity to iodine or iodinated contrast agents.
  3. Patients with serious thyroid disease (goiter, hyperthyroidism, etc.)
  4. Patients with serious cardiopathy (NYHA functional class IV heart failure as described in Appendix 5, shock, cyanosis, peripheral circulatory insufficiency, ventricular tachycardia, ventricular fibrillation, or complete atrioventricular block)
  5. Patients with serious hepatopathy (symptoms of liver failure [fulminant hepatitis] such as a disturbance of consciousness corresponding to grade 3 in the Criteria for Grading Adverse Drug Reactions of Medicinal Products in Appendix 5).
  6. Patients with moderate or serious nephropathy (acute or chronic renal failure, hydronephrosis, nephrotic syndrome, or uremia with serum creatinine levels of 2.0 mg/dL or above, corresponding to grade 2 or above in the Criteria for Grading Adverse Drug Reactions of Medicinal Products in Appendix 5).
  7. Patients with bronchial asthma
  8. Patients with acute pancreatitis
  9. Patients with macroglobulinemia
  10. Patients with multiple myeloma
  11. Patients with tetany
  12. Patients with pheochromocytoma or who are suspected to be pheochromocytoma
  13. Women of pregnant, childbearing potential, or lactating
  14. Patients with a history of hypersensitivity to drug(s)
  15. Patients with hypertension under medication
  16. Patients with diabetes under medication
  17. Patients with serious illness myasthenia
  18. Patients judged to be ineligible for study entry by an investigator or subinvestigator for any other reasons

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Efficacy
Contrast enhancement effect in the early arterial phase
Safety
Warming sensation and vascular pain

SECONDARY OUTCOMES:
Efficacy
Contrast enhancement effect in the portal phase
Safety and arterial, portal venous and liver parenchymal CT values (HU)
Symptoms and signs（excluding warming sensation and vascular pain ）, and life signs (blood pressure, pulse), etc., and laboratory tests (hematology, serum chemistry) conducted before and after administration of the investigational agent

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Tazawa, Study Director — Eisai Co., Ltd - Development Clinical Research Department. Clinical Research Center
Locations (2):
- Japan (2):
  - Kumamoto, Kumamoto
  - Suita, Osaka